CLINICAL TRIAL: NCT06920186
Title: Comparison of the Benefit of Peripheral Nerve Quadri-block Versus Adductor Canal Block + Surgical Infiltration in Total Knee Arthroplasty
Brief Title: Infiltration or Nerve Blocks in Addition to Adductor Canal Block
Acronym: INCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: COS-RGDS-2024-06-006-P-ELMALEH; 2024-A02496-41 (Other: N° ID-RCB (ANSM))
Record Dates: First submitted 2025-03-24; First posted 2025-04-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gonarthrosis; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Analgesia

STUDY DESIGN:
Intervention Model Description: Category 2 Research Involving the Human Person (RIPH 2) :
  Multi-center (2 sites), prospective, double-blind randomized, open-label study of two parallel groups of patients undergoing total knee arthroplasty according to locoregional analgesia (LRA) protocol :
  * Group 1: Real adductor canal block + surgical infiltration and sham of femoro-cutaneous block + obturator block + IPACK block with physiological serum
  * Group 2: Real adductor canal block + femoro-cutaneous block + obturator block + IPACK block and sham of surgical infiltration with physiological serum
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 of local analgesia protocol (PROSPECT recommandations) (Sham Comparator): Locoregional analgesia (LRA) protocol n°1 : adductor canal block + surgical infiltration (PROSPECT recommendations)
  Interventions: Procedure: Analgesia
- Group 2 of local analgesia protocol (quadri-peripheral nerve block ) (Experimental): Locoregional analgesia (LRA) protocol n° 2 : adductor canal block + femoral-cutaneous block + obturator block + IPACK block
  Interventions: Procedure: Analgesia

INTERVENTIONS:
Procedure: Analgesia — 1- Real Adductor canal block + surgical infiltration and sham of femoro-cutaneous block + obturator block + IPACK block with physiological serum
  Arms: Group 1 of local analgesia protocol (PROSPECT recommandations)
Procedure: Analgesia — 2- Real Adductor canal block + femoral-cutaneous block + obturator block + IPACK block and sham of surgical infiltration with physiological serum
  Arms: Group 2 of local analgesia protocol (quadri-peripheral nerve block )

SUMMARY:
The aim of this study is to evaluate the analgesic efficacy of this quadruple sensory block compared with the currently recommended procedure (adductor canal block + infiltration).

DETAILED DESCRIPTION:
In addition to the adductor canal block, this quadruple block incorporates :

1. the block of the lateral cutaneous nerve of the thigh (or femoral-cutaneous nerve), which is a collateral sensory branch of the posterior part of the lumbar plexus.
2. IPACK (Infiltration between Popliteal Artery and Capsule of Knee), designed as a motor-sparing technique (targeting the sensory articular branches of the sciatic nerve and avoiding the motor branches of the tibial and fibular nerves), is particularly effective on posterior pain.
3. obturator nerve block, a mixed nerve originating from the anterior part of the lumbar plexus. It divides into two branches: anterior, which innervates the adductor longus, adductor brevis and gracilis muscles, and posterior, which innervates the medial part of the knee joint and the posteromedial part of the thigh. It provides sensitivity to the medial aspect of the thigh.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female
* Patient with signed consent to participate in the study,
* Patient with uni or bilateral primary gonarthrosis
* Indication for total knee arthroplasty.

Exclusion Criteria:

* History of knee fracture, arthroplasty or osteotomy
* Known or unknown contraindication to ALR or locoregional anesthesia products
* Neurological disease, stroke sequelae
* Mental deficiency or any other reason that may hinder understanding or strict application of the protocol
* Patient not affiliated to the French social security system
* Patient under court protection, guardianship or curatorship
* Pregnant or potentially pregnant women (women of childbearing age without effective contraception)
* Patient already included in another therapeutic study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Patient's recovery at H24 as after surgery assessed by the QoR-15 (Quality of Recovery) questionnaire score | From enrollement to the last H24 after surgery
  The QoR-15 score at H24 after surgery was compared between the two groups for primary endpoint analysis.
  The QoR-15 accurately measures postoperative recovery by focusing on 5 key domains: pain, physical comfort, physical independence, psychological support and emotional state. Each item is rated from 0 (unfavorable) to 10 (favorable), with an overall score corresponding to the sum of the score obtained for each item, i.e. a score from 0 (no recovery) to 150 (full recovery).

SECONDARY OUTCOMES:
Knee functional assessment | Hour 0
  Functional assessment of the knee with KOOS JR questionnaire
Post operative pain | Hour 2
  Pain measured with a simple numeric scale
Post operative pain | Hour 6
  Pain measured with a simple numeric scale
Post operative pain | Hour 12
  Pain measured with a simple numeric scale
First ambulation | Hour 12
  time between end of intervention and first ambulation
Post operative pain | Hour 24
  Pain measured with a simple numeric scale
Joint range of both knees | Hour 24
  Measurement of the joint range of both knees
First ambulation | Hour 24
  time between end of intervention and first ambulation
Post operative pain | Hour 48
  Pain measured with a simple numeric scale
Quality of recovery | Hour 48
  Quality of recovery measured with QoR 15 questionnaire
Opioid drug use | Hour 48
  Opioid drug use evaluation
Non-opioid drug use | Hour 48
  Non-opioid drug use evaluation
Joint range of both knees | Hour 48
  Measurement of the joint range of both knees
First ambulation | Hour 48
  time between end of intervention and first ambulation
Length of stay in the post-intervention monitoring room | Hour 48
  Length of stay in the post-intervention monitoring room
Post operative pain | Month 1
  Pain measured with a simple numeric scale
Joint range of both knees | Month 1
  Measurement of the joint range of both knees
Length of hospitalisation | Month 1
  Length of hospitalisation
Return to patient usual activities | Month 1
  Time taken for the patient to return to their usual activities
Drug tolerance | Month 1
  Drug tolerance
Patient comfort | Hour 1
  Patient comfort during loco-regional anesthesia
Knee functional assessment | Month 1
  Functional assessment of the knee with KOOS JR questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Privé Claude Galien, Quincy-sous-Sénart
  - Clinique des Côtes du Rhône, Roussillon

IPD SHARING:
Plan to Share IPD: No